CLINICAL TRIAL: NCT05502848
Title: The Effect of Intervention and Mechanism of Internet Cognitive Behavioral Therapy on Chronic Itching in Patients With Atopic Dermatitis
Brief Title: The Effect of Intervention and Mechanism of ICBT on Chronic Itching in Patients With Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2209090555263
Record Dates: First submitted 2022-08-01; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Internet Cognitive Behavioral Therapy; Chronic Itching; Functional MRI
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AD patients treated with ICBT (Experimental)
  Interventions: Behavioral: Internet Cognitive Behavior Therapy
- AD patients receiving regular treatment (No Intervention)
- Healthy Controls (No Intervention)

INTERVENTIONS:
Behavioral: Internet Cognitive Behavior Therapy — ICBT helps change patterns of thinking (cognitions) and behaviors of psychological distress, including relaxation, stress management, while using ICBT can increase personal tolerance for negative thoughts and negative emotions, help patients reduce negative perception of the disease due to long-term recurrent itching, and break the vicious cycle
  Arms: AD patients treated with ICBT

SUMMARY:
Objectives: The study subjects were 180 healthy people from the dermatology clinic of Xiangya Hospital of Central South University and the surroundingcommunity, including 120 AD patients (60 in the ICBT treatment group and 60 in the control group) and 60 healthy controls.

Methodology: After obtaining the informed consent of the subjects, the general condition and clinical symptoms of the subjects were assessed, the cognitive and psychological characteristics of the subjects who met the inclusion were assessed, multimodality MRI was scanned and blood and saliva samples were collected. The same assessments and data collection were performed with healthy controls matched for age, sex, and years of education in the AD patient group. AD patients were randomly assigned to the ICBT intervention group (n = 60) by a random number table and immediately started ICBT adjuvant therapy, or the control group (n = 60) for conventional therapy. Clinical symptoms and cognitive psychological characteristics of AD patients were assessed at the end of 2 weeks, 4 weeks, 8 weeks, 6 months and 12 months of ICBT treatment, and cognitive behavioral task measurements, multimodality magnetic resonance scans, blood and saliva samples will be performed again at the follow-up time point at the end of 6 months. Healthy controls (60) will also undergo a full set of follow-up assessments again after 6 months.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common chronic inflammatory skin disease accompanied by severe itching, leading to poor patient-reported satisfaction. Previous studies have found a mutually reinforcing relationship between stress, depression, anxiety and itching in AD, which is mediated by cognitive dysfunction. Patients with AD show elevated activation in the key regions of cognitive control network, such as anterior cingulate cortex and dorsolateral prefrontal cortex, when facing itching stimulus, which are positively associated with the severity of itching. Based on these findings, we propose a hypothesis that "dysfunction of cognitive control network may underlie the increased sensitivity to itching in AD". To test the hypothesis, we will conduct a randomized controlled study on the effectiveness of Internet cognitive behavior therapy (ICBT) for AD. Using the multi-modal magnetic resonance imaging technology, we will compare the brain imaging characteristics in AD patients before and after treatment with ICBT. We will further investigate the factors associated with response to ICBT treatment and the underlying mechanisms of the treatment effect of ICBT, expecting to improve long-term treatment outcomes of AD.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria of AD
* more than moderate AD symptoms, with patient-oriented eczema measurement score (POEM) ≥ 8 points, atopic dermatitis score (SCORAD) objective signs score > 15 points
* aged 18-45 years
* right-handed
* education years ≥ 6 years and access to the Internet
* patients must stop all immunosuppressive drugs at least 10 days before the study to avoid potential itching inhibition
* voluntarily participate in this study, and have fully understood the purpose, methods, procedures, possible discomfort and risks of the experiment, and signed informed consent.

Exclusion Criteria:

* current or previous severe physical and neurological diseases
* chronic oral benzodiazepines and other drugs
* recent or ongoing psychotherapy
* psoriasis
* recent ultraviolet therapy or immunosuppressive drug therapy for AD
* patients at serious risk of suicide
* claustrophobia or metal implants in the body. (Considering the effect of age on MRI results, only patients aged 18-45 years were included in this study. After enrollment, conventional treatment such as topical glucocorticoids was not affected by this study, but the two groups were matched in the selection of conventional treatment drugs. On this basis, patients were randomly divided into ICBT intervention group or conventional treatment control group)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Patient Oriented Eczema Measure(POEM) | Baseline and Week 2;4;8 and Month 6;12
  Patient Oriented Eczema Measure (POEM) is divided into 7 questions, with a total score of 28 points, and treatment response is defined as a reduction of POEM of greater than 4 points
Change from Baseline on the Scoring Atopic Dermatitis Index(SCORAD) | Baseline and Week 2;4;8 and Month 6;12
  Scoring Atopic Dermatitis Index (SCORAD), which consists of objective signs (lesion area, lesion severity) and subjective symptoms as well as a visual analogue scale assessing pruritus and sleep impact.
Change from Baseline on scratching times | Baseline and Week 2;4;8 and Month 6;12
Change from Baseline on the Itchy Quality of Life(ItchyQoL) | Baseline and Month 6
  Itchy Quality of Life (Itchy QoL): assess the impact of pruritus symptoms on quality of life. The Chinese version of Itchy Quality of Life (QOL) consists of 22 items, including three dimensions of symptoms, mood and functional activities, with good reliability and validity
Change from Baseline on structural MRI (3D; DTI) and functional MRI (resting state; task state) | Baseline and Month 6
  MRI data were acquired on a Siemens scanner using a 64-channel head coil，We used structural MRI to measure voxel-base morphometry analysis of brain regions as well as changes in DTI connectivity activity. We will compare structural and functional magnetic resonance differences between AD and healthy controls, structural magnetic resonance and functional magnetic resonance differences between AD after 6 months of ICBT therapy, AD control and baseline, and differences between AD and healthy controls after 6 months

SECONDARY OUTCOMES:
Change from Baseline on the 9-item Patient Health Questionnaire(PHQ-9) | Baseline and Week 2;4;8 and Month 6;12
  9-item Patient Health Questionnaire (PHQ-9): used to assess severity of depression
Change from Baseline on the Generalized Anxiety Disorder-7(GAD-7) | Baseline and Week 2;4;8 and Month 6;12
  7-item Generalized Anxiety Disorder-7 (GAD-7): used to assess anxiety severity in subjects
Change from Baseline on the Athens Insomnia ScaleL(AIS) | Baseline and Month 6
  Athens Insomnia ScaleL (AIS): It is used to evaluate the sleep status of subjects
Change from Baseline on the Dysfunctional Attitude Scale(DAS) | Baseline and Month 6
  Dysfunctional Attitude Scale (DAS): a total of 40 items, assess the subjective cognitive attitude of subjects, assess the subjective cognitive attitude of subjects to self, external events and negative perceptions of the future, including vulnerability, attraction and rejection, perfection, compulsion, praise seeking, dependence, autonomy attitude and cognitive philosophy. The higher the score, the stronger the negative understanding of patients.
Change from Baseline on the blood samples | Baseline and Month 6
  Cortisol level (ng/ml), ATP(nmmol/L), highly sensitive C-reactive protein (hs-CRP), Monocyte Chemoattractant Protein 1 (MCP1), Type 2 inflammation: interleukins (IL)-4, 5, 13, 31, Type 1 inflammation: Tumor necrosis factor(TNF), Interferon(IFN)γ, Type 17-22 inflammation: IL-12, IL-23, IL-17a, IL-22, Innate inflammation: thymic stromal lymphopoietin(TSLP), IL-25, IL-33, IL-1b, IL-1a, IL-18
Change from Baseline on Attention Network Test (ANT) | Baseline and Month 6
  Attention Network Test (ANT) experimental paradigm: This paradigm can effectively measure the efficiency of three core components of attention network (alerting, orienting and executive function).
Change from Baseline on THINC-integrated tool | Baseline and Month 6
  THINC-it tool (THINC - integrated tool) cognitive test: It is a digital cognitive assessment screening tool that integrates a series of assessments: patients with cognitive deficits ask, this questionnaire is a subjective assessment questionnaire of patients' cognitive function.
Change from Baseline on the Chinese Perceived Stress Scale (CPSS) | Baseline and Month 6
  The Chinese Perceived Stress Scale (CPSS) assesses individual stress in subjects. This scale asks how you have been feeling and thinking in the last month, with higher scores indicating greater stress

IPD SHARING:
Plan to Share IPD: No